CLINICAL TRIAL: NCT01916902
Title: Effect of Pretreatment With Ticagrelor on Residual Thrombus After Percutaneous Coronary Intervention (PCI) in Patients Presenting With Acute Coronary Syndrome in Comparison With Delayed Treatment at the Time of PCI: an Optical Coherence Tomography Study
Brief Title: Effect of Pretreatment With Ticagrelor on Residual Thrombus After PCI in Patients Presenting With ACS in Comparison With Delayed Treatment at the Time of PCI: an OCT Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Despite a large number of patients screened, very few met eligibility guidelines.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2013P001322
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Optical Coherence Tomography; Ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Ticagrelor- Delayed Administration (Active Comparator): Subjects receive 180 mg of ticagrelor during cardiac catheterization after diagnostic angiography and prior to stenting. OCT is performed prior to and after coronary artery stenting.
  Interventions: Drug: Ticagrelor- Delayed Administration; Procedure: Optical Coherence Tomography
- Ticagrelor- Immediate Administration (Active Comparator): Subjects receive 180 mg of ticagrelor immediately after study enrollment. OCT is performed prior to and after coronary artery stenting.
  Interventions: Drug: Ticagrelor- Immediate Administration; Procedure: Optical Coherence Tomography

INTERVENTIONS:
Drug: Ticagrelor- Delayed Administration — Subjects are randomized to receive ticagrelor immediately after enrollment versus at the time of cardiac catheterization. OCT is performed prior to and after coronary artery stenting.
  Arms: Ticagrelor- Delayed Administration
Drug: Ticagrelor- Immediate Administration — Subjects are randomized to receive ticagrelor immediately after enrollment versus at the time of cardiac catheterization. OCT is performed prior to and after coronary artery stenting.
  Arms: Ticagrelor- Immediate Administration
Procedure: Optical Coherence Tomography

SUMMARY:
Subjects presenting with probable acute coronary syndromes scheduled for cardiac catheterization will be enrolled in this study. Consented subjects will be randomized to receive ticagrelor started with a loading dose immediately after enrollment versus receiving a loading dose of ticagrelor during cardiac catheterization after diagnostic angiography but prior to stenting. Optical coherence tomography (OCT) will be performed after stenting and the volume of thrombus within the new stent will be measured and compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

Patient Characteristics:

1. Males and non-pregnant females > or equal to 18 and < or equal to 79 years of age presenting with suspected acute coronary syndrome (unstable angina or NSTEMI)
2. Patients likely to be scheduled to undergo coronary angiography with possible percutaneous coronary intervention (PCI)

Lesion Characteristics on Diagnostic Coronary Angiography:

1. De novo lesions in native coronary arteries found by diagnostic coronary angiography
2. Angiographic stenosis <100%
3. Reference vessel diameter 2.5 mm - 4.0 mm by visual estimation

Exclusion Criteria:

Patient Specific Exclusion Criteria:

1. Subjects who are unable or unwilling to sign the informed consent form.
2. Subjects being treated with anti-platelet medications other than aspirin prior to diagnostic catheterization including glycoprotein IIb/IIIa inhibitors.
3. Subjects with serious co-morbid conditions that in judgment of the investigator preclude inclusion in this study
4. Subjects with NYHA class III or IV heart failure or known left ventricular ejection fraction < 30%.
5. Subjects with an ST elevation myocardial infarction.
6. Subjects with hemodynamic or electrical instability (including shock).
7. Subjects diagnosed with severe, non-catheter-related coronary artery spasm.
8. Subjects who are or may be pregnant.
9. Subjects with known allergies to contrast media.
10. Subjects with eGFR < 60 ml/min/1.73m2.
11. Subjects currently taking oral anticoagulants with an absolute contraindication to discontinuation of anticoagulation.
12. History of TIA or stroke < 6 months.
13. History of hemorrhagic stroke.
14. Hepatic insufficiency defined as liver cirrhosis, AST/ALT/Alkaline Phosphatase greater than 3 times the upper limit of normal or hyperbilirubinemia.
15. Cardiac catheterization scheduled within 4 hours of randomization or more then 72 hours after randomization.

Lesion Specific Exclusion Criteria. These exclusion criteria apply to the target lesion to be imaged by OCT.

1. Lesions located in the left main coronary artery
2. Lesions that are heavily calcified
3. Lesions where OCT cannot be performed due to technical difficulties
4. Other lesions that the investigator deems inappropriate for the procedure such as sites with excessive tortuosity or low flow by TIMI grade.
5. Lesions in saphenous vein grafts or arterial conduits.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Total thrombus burden as measured by the volume of in-stent thrombus quantified by planimetry. | Thrombus burden will be measured at the end of the coronary artery stenting procedure.
  The total thrombus burden measured on OCT images will be assessed. The volume of in-stent thrombus will be quantified by planimetry.

SECONDARY OUTCOMES:
PRI (platelet reactivity index) as measured bu the PLT-VASP assay. | PRI iwill be measured at the time of OCT image acquisition.
  The extent of platelet inhibition will be measured by PLT-VASP and VerifyNow P2Y12 assays.
P2Y12 Reaction Units as measured by the VerifyNow P2Y12 assay. | P2Y12 will be measured at the time of OCT image acquisition.
  The extent of platelet inhibition will be measured by PLT-VASP and VerifyNow P2Y12 assays.

OTHER OUTCOMES:
PCI-related myocardial infarction (MI) | PCI-related MI will be assesed within 24 hours after the end of the coronary artery stenting procedure.
  PCI related myocardial infarction is defined by the third Universal definition of myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States